CLINICAL TRIAL: NCT01359449
Title: Safety and Immunogenicity of Two Doses of Menactra® (Meningococcal [Groups A, C, Y, and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) or One Dose of Monovalent Meningococcal Group C Conjugate Vaccine Administered Concomitantly With Routine Immunizations Between 12 and 18 Months of Age in Canada
Brief Title: Study of Two Doses of Menactra® or One Dose of Monovalent Meningococcal Group C Vaccine With Routine Immunizations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA73; U1111-1117-7073 (Other: WHO)
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection; Menactra®; MenC
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menactra® Vaccine Group (Experimental): Meningococcal vaccine naive participants will receive Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate vaccine (Menactra®) at 12 months of age and at 18 months of age concomitantly with routine vaccines administered as per provincial schedule
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate: Menactra®
- Menjugate® Vaccine Group (Active Comparator): Meningococcal vaccine naive participants will receive MenC vaccine (Menjugate) given concomitantly at 12 months of age with routine vaccines administered as per provincial schedule.
  Interventions: Biological: Meningococcal Group C Conjugate vaccine: MenC

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate: Menactra® — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Vaccine Group
Biological: Meningococcal Group C Conjugate vaccine: MenC — 0.5 mL, Intramuscular
  Other Names: Menjugate; MenC
  Arms: Menjugate® Vaccine Group

SUMMARY:
The purpose for this study is to demonstrate the safety and immunogenicity of two doses of Menactra® administered between 12 and 18 months of age and concomitantly with routine immunization with two different provincial schedule

Primary Objectives:

* To describe the immunogenicity of Menactra® administered concomitantly with routine immunizations at 12 and 18 months in naïve or Menjugate-primed (MenC-primed) infants (measured by serum bactericidal assay using baby rabbit complement [SBA-BR])
* To describe the immunogenicity of MenC administered concomitantly with routine immunizations at 12 months of age (measured by SBA-BR)

Secondary Objectives:

Safety

* To describe the safety profile of Menactra® and MenC vaccines after each dose when given concomitantly with routine immunization.

Immunogenicity

* To describe the immunogenicity of both vaccines using serum bactericidal assay using human complement [SBA-HC]
* To describe the immunogenicity of Pediacel administered at 18 months.

DETAILED DESCRIPTION:
Participants depending on their groups will receive either two doses of Menactra vaccine concomitantly with the routinely recommended vaccines or one dose of MenC vaccine concomitantly with the routinely recommended vaccines and will be monitored for safety and immunogenicity. The duration of each subject's participation in the trial will be approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 months (365 to 400 days) on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Informed consent form has been signed and dated by the parent(s) or other legally authorized representative
* Subject and parent/legal representative are able to attend all scheduled visits and to comply with all trial procedures
* Group 1: Subject has received 3 primary vaccination doses of Pediacel as per routine immunization schedule
* Group 3: Subject has received two doses of MenC vaccine at approximately 2 and 4 months of age as per Alberta immunization schedule.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for influenza vaccination(s), which may be received at least two weeks before study vaccines
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Previous vaccination against Meningococcal disease OR
* Subject has previously received only one dose of MenC vaccine, or more than two doses of MenC vaccine, or two doses of MenC vaccine with the most recent dose received in the past 6 months
* Receipt of blood or blood-derived products in the past 3 months which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal or maternal seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, as reported by the parent/legal representative
* History of documented invasive meningococcal disease
* At high risk for meningococcal disease during the trial
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* History of contraindication to receipt of pertussis-containing vaccine
* Thrombocytopenia, as reported by the parent/legal representative, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* History of seizures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* History of Guillain-Barré Syndrome.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Dierctor, Study Director — Sanofi Pasteur SA
Locations (1):
- Pierrefonds, Quebec, Canada

REFERENCES:
- [Result] Noya F, McCormack D, Reynolds DL, Neame D, Oster P. Safety and immunogenicity of two doses of quadrivalent meningococcal conjugate vaccine or one dose of meningococcal group C conjugate vaccine, both administered concomitantly with routine immunization to 12- to 18-month-old children. Can J Infect Dis Med Microbiol. 2014 Jul;25(4):211-6. doi: 10.1155/2014/237560. PMID 25285126
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 19 May 2011 through 14 September 2011 in one clinic site in Canada.
Pre-assignment Details: A total of 123 participants that met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Menactra® Vaccine Group: Participants received one dose of Menactra® vaccine at 12 months of age and a second dose on Menactra® vaccine at 18 months of age concomitantly with routine vaccines administered as per provincial schedule (including the 4th dose of Pediacel® at 18 months of age)
- Menjugate® Vaccine Group: Participants received Menjugate® vaccine given concomitantly at 12 months of age with routine vaccines administered as per provincial schedule.
Period: Overall Study
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Started | 61 | 62
Completed | 57 | 58
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 62 | 123
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.4 (0.3) | 12.4 (0.3) | 12.4 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 27 | 29 | 56
Region of Enrollment [Number; unit: Participants]
  Canada | 61 | 62 | 123

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Serum Bovine Albumin Baby Rabbit Titers Following Vaccination With Either One Dose of Menactra® Vaccine at 12 and 18 Months of Age, Respectively, or One Single Dose of Menjugate® Vaccine at 12 Months of Age.
Description: Immunogenicity tests were performed at 19 months of age in Menactra Vaccine Group after Menactra® vaccination and performed at 13 months and 19 months of age in the Menjugate Vaccine Group after Menjugate® vaccination
Time Frame: 28 days post-vaccination
Population: Geometric Mean Titers of Serum Bovine Albumin Baby Rabbit titers were determined in the per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 55 | 62
Titers
  Serogroup A (at age13 months, N = 0, 60) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 4.34 [3.69 to 5.10]
  Serogroup A (at age 19 months, N = 51, 58) | 1740 [1301 to 2327] | 4.35 [3.76 to 5.03]
  Serogroup C (at age 13 months, N = 0, 60) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 71.0 [39.3 to 128]
  Serogroup C (at age 19 months, N = 51, 58) | 957 [594 to 1540] | 11.0 [6.75 to 18.1]
  Serogroup Y (at age 13 months, N = 0, 60) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 31.3 [19.6 to 50.0]
  Serogroup Y (at age 19 months, N = 51, 58) | 719 [553 to 935] | 67.1 [38.4 to 117]
  Serogroup W-135 (at age 13 months, N = 0, 60) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 5.28 [4.13 to 6.74]
  Serogroup W-135 (at age 19 months, N = 51, 58) | 970 [686 to 1371] | 7.36 [5.24 to 10.3]

2. Primary Outcome: Number of Participants With Serum Bovine Albumin Baby Rabbit Titers of ≥ 1:8 Following Vaccination With Either a Dose of Menactra Vaccine at 12 and 18 Months of Age, Respectively, or One Single Dose of Menjugate® Vaccine at 12 Months of Age.
Description: as for outcome 1
Time Frame: 28 days post-vaccination
Population: Immunogenicity using Serum Bovine Albumin Baby Rabbit titers were determined in the per-protocol population
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 55 | 62
Participants
  Serogroup A (at age 13 months; N = 0, 60) | NA — Data not determined for this group at this time point as per protocol. | 1 [0 to 0]
  Serogroup A (at age 19 months; N = 51, 58) | 51 | 2 [0 to 0]
  Serogroup C (at age 13 months; N = 0, 60) | NA — Data not determined for this group at this time point as per protocol. | 40 [0 to 0]
  Serogroup C (at age 19 months; N = 51, 58) | 49 | 15 [0 to 0]
  Serogroup Y (at age 13 months; N = 0, 60) | NA — Data not determined for this group at this time point as per protocol. | 36 [0 to 0]
  Serogroup Y (at age 19 months; N = 51, 58) | 51 | 39 [0 to 0]
  Serogroup W-135 (at age 13 months; N = 0, 60) | NA — Data not determined for this group at this time point as per protocol. | 5 [0 to 0]
  Serogroup W-135 (at age 19 months; N = 51, 58) | 50 | 11 [0 to 0]

3. Secondary Outcome: Geometric Mean Titers of Serum Bovine Albumin Human Complement Titers Following Vaccination With Either One Dose of Menactra® Vaccine at 12 and 18 Months of Age, Respectively, or One Single Dose of Menjugate® Vaccine at 12 Months of Age.
Description: as for outcome 1
Time Frame: 28 days post-vaccination
Population: Geometric Mean Titers of Serum Bovine Albumin Human Complement titers were determined in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 55 | 62
Titers
  Serogroup A (at age 13 months, N = 0, 44) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 2.23 [2.04 to 2.44]
  Serogroup A (at age 19 months, N = 49, 48) | 71.7 [48.2 to 107] | 2.21 [2.00 to 2.45]
  Serogroup C (at age 13 months, N = 0, 50) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 17.4 [11.6 to 26.1]
  Serogroup C (at age 19 months, N = 49, 53) | 219 [152 to 315] | 6.93 [4.53 to 10.6]
  Serogroup Y (at age 13 months, N = 0, 45) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 2.00 [2.0 to 2.0]
  Serogroup Y (at age 19 months, N = 49, 53) | 299 [222 to 403] | 2.14 [1.98 to 2.31]
  Serogroup W-135 (at age 13 months, N = 0, 45) | NA [NA to NA] — Data not determined for this group at this time point as per protocol. | 2.06 [1.97 to 2.15]
  Serogroup W-135 (at age 19 months, N = 49, 50) | 207 [146 to 295] | 2.17 [2.01 to 2.34]

4. Secondary Outcome: Number of Participants With Serum Bovine Albumin Human Complement Titers of ≥ 1:8 Following Vaccination With Either a Dose of Menactra® Vaccine at 12 and 18 Months of Age, Respectively, or One Single Dose of Menjugate® Vaccine at 12 Months of Age.
Description: as for outcome 1
Time Frame: 28 days post-vaccination
Population: Immunogenicity using Serum Bovine Albumin Human Complement titers were determined in the per-protocol population
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 55 | 62
Participants
  Serogroup A (at age 13 months; N = 0, 44) | NA — Data not determined for this group at this time point as per protocol. | 1 [0 to 0]
  Serogroup A (at age 19 months; N = 49, 48) | 48 | 1 [0 to 0]
  Serogroup C (at age 13 months; N = 0, 50) | NA — Data not determined for this group at this time point as per protocol. | 39 [0 to 0]
  Serogroup C (at age 19 months; N = 49, 53) | 49 | 21 [0 to 0]
  Serogroup Y (at age 13 months; N = 0, 45) | NA — Data not determined for this group at this time point as per protocol. | 0 [0 to 0]
  Serogroup Y (at age 19 months; N = 49, 53) | 49 | 2 [0 to 0]
  Serogroup W-135 (at age 13 months; N = 0, 45) | NA — Data not determined for this group at this time point as per protocol. | 0 [0 to 0]
  Serogroup W-135 (at age 19 months; N = 49, 50) | 48 | 1 [0 to 0]

5. Secondary Outcome: Geometric Mean Titers of Antibodies to Pediacel® Vaccine Antigens in Participants That Received a Dose of Menactra® at 12 and 18 Months of Age, Respectively, and a Booster Dose of Pediacel® Vaccine at 18 Months of Age.
Description: Immunogenicity tests were performed at 18 and 19 months of age, respectively, before and after Pediacel® vaccination in the Menactra vaccine group
Time Frame: 28 days post-vaccination
Population: Geometric Mean Titers of of Pediacel vaccine antigens were determined in the per-protocol population of the Menactra® vaccine group.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 51 | 62
Titers
  Diphtheria (at age 18 months; N = 46, 0) | 0.420 [0.283 to 0.622] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Diphtheria (at age 19 months; N = 46, 0) | 7.81 [6.03 to 10.1] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Tetanus (at age 18 months; N = 44, 0) | 0.485 [0.365 to 0.644] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Tetanus (at age 19 months; N = 47, 0) | 8.71 [7.02 to 10.8] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  PRP (at age 18 months; N = 44, 0) | 0.500 [0.306 to 0.818] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  PRP (at age 19 months; N = 46, 0) | 46.3 [32.2 to 66.4] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 1 (at age 18 months; N = 45, 0) | 138 [95.2 to 201] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 1 (at age 19 months; N = 46, 0) | 4552 [3436 to 6029] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 2 (at age 18 months; N = 39, 0) | 203 [127 to 324] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 2 (at age 19 months; N = 46, 0) | 6889 [5250 to 9039] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 3 (at age 18 months; N = 38, 0) | 133 [84.2 to 209] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Polio Type 3 (at age 19 months; N = 45, 0) | 5322 [3705 to 7645] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Pertussis Toxoid (at age 18 months; N = 45, 0) | 8.61 [6.39 to 11.6] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Pertussis Toxoid (at age 19 months; N = 47, 0) | 162 [132 to 199] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Filamentous hemagglutinin (age 18 months; N=45, 0) | 19.9 [14.1 to 28.2] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Filamentous hemagglutinin (age 19 months; N=47, 0) | 239 [182 to 315] | NA [NA to NA] — Participants in this group did not receive Pediacel vaccine in this study.
  Pertactin (at age 18 months; N = 44, 0) | 8.45 [6.46 to 11.0] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Pertactin (at age 19 months; N = 45, 0) | 123 [90.7 to 165] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Fimbriae types 2 and 3 (age 18 months; N = 45, 0) | 35.7 [26.4 to 48.3] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.
  Fimbriae types 2 and 3 (age 19 months; N = 45, 0) | 622 [425 to 911] | NA [NA to NA] — Participants in this group did not receive Pediacel® vaccine in this study.

6. Secondary Outcome: Summary of Participants With Booster Response for Pediacel® Vaccine Antigens After Vaccination With Pediacel® Vaccine (Menactra Vaccine Group)
Description: Pediacel vaccine administered only to the Menactra Vaccine Group. Booster response was defined as subjects with pre-dose titers < 4xLLOQ and have a 4-fold rise rate; or subjects with pre-dose titers ≥ 4xLLOQ and have a 2-fold rise rate
Time Frame: 28 days post-vaccination
Population: Pediacel® vaccine antigen booster responses were determined in the per-protocol population of the Menactra® vaccine group
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 51 | 62
Participants
  Pertussis toxoid (N = 44, 0) | 44 | NA — Participants in this group did not receive Pediacel® vaccine in this study.
  Filamentous hemagglutinin (N = 44, 0) | 43 | NA — Participants in this group did not receive Pediacel® vaccine in this study.
  Pertactin (N = 41, 0) | 38 | NA — Participants in this group did not receive Pediacel® vaccine in this study.
  Fimbriae types 2 and 3 (N = 42, 0) | 42 | NA — Participants in this group did not receive Pediacel® vaccine in this study.

7. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Following Vaccination With Either a Dose of Menactra Vaccine at 12 and 18 Months of Age, Respectively, or One Single Dose of Menjugate Vaccine at 12 Months of Age
Description: Solicited Injection site: Tenderness, Erythema and Swelling: Solicited Systemic: Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability.
  Grade 3 reactions defined as: Tenderness - Cries when injected limb is moved, or the movement of the injected limb is reduced; Erythema and Swelling - ≥ 50 mm; Fever - > 39.5°C; Vomiting - ≥ 6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal - > 3 hours; Drowsiness - Sleeping most of the time or difficult to wake up; Appetite lost - Refuses ≥ 3 feeds/meals or refuses most feeds/meals, and Irritability - Inconsolable.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all enrolled and vaccinated participants, intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 60 | 62
Participants
  Any injection site Tenderness | 21 | 21 [0 to 0]
  Grade 3 injection site Tenderness | 0 | 0 [0 to 0]
  Any injection site Erythema | 26 | 23 [0 to 0]
  Grade 3 injection site Erythema | 0 | 0 [0 to 0]
  Any injection site Swelling | 9 | 8 [0 to 0]
  Grade 3 injection site Swelling | 0 | 0 [0 to 0]
  Any Fever | 30 | 18 [0 to 0]
  Grade 3 Fever | 1 | 0 [0 to 0]
  Any Vomiting | 5 | 7 [0 to 0]
  Grade 3 Vomiting | 0 | 0 [0 to 0]
  Any Crying abnormal | 25 | 22 [0 to 0]
  Grade 3 Crying abnormal | 0 | 0 [0 to 0]
  Any Drowsiness | 22 | 12 [0 to 0]
  Grade 3 Drowsiness | 0 | 0 [0 to 0]
  Any Appetite lost | 28 | 24 [0 to 0]
  Grade 3 Appetite lost | 0 | 0 [0 to 0]
  Any Irritability | 43 | 40 [0 to 0]
  Grade 3 Irritability | 1 | 1 [0 to 0]

8. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Following Vaccination With a Second Dose of Menactra Vaccine at 18 Months of Age
Description: as for outcome 7
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all enrolled and vaccinated participants in the Menactra vaccine group, intent to treat population
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 60 | 62
Participants
  Any injection site Tenderness | 30 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 injection site Tenderness | 2 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any injection site Erythema | 19 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 injection site Erythema | 1 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any injection site Swelling | 11 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 injection site Swelling | 0 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Fever | 21 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Fever | 3 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Vomiting | 6 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Vomiting | 1 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Crying abnormal | 25 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Crying abnormal | 1 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Drowsiness | 20 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Drowsiness | 1 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Appetite lost | 32 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Appetite lost | 1 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Any Irritability | 40 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.
  Grade 3 Irritability | 2 | NA [0 to 0] — Participants in this group did not receive a second dose of a meningococcal vaccine in this study.

9. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Following Any of the Study Vaccination
Description: Solicited Injection site: Tenderness, Erythema and Swelling: Solicited Systemic: Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability
Time Frame: Day 0 up to Day 7 post-vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Number analyzed (Participants) | 60 | 62
Participants
  Any injection site Tenderness | 36 | 21 [0 to 0]
  Any injection site Erythema | 32 | 23 [0 to 0]
  Any injection site Swelling | 18 | 8 [0 to 0]
  Any Fever | 44 | 18 [0 to 0]
  Any Vomiting | 10 | 7 [0 to 0]
  Any Crying abnormal | 31 | 22 [0 to 0]
  Any Drowsiness | 31 | 12 [0 to 0]
  Any Appetite lost | 45 | 24 [0 to 0]
  Any Irritability | 50 | 40 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Day 0 (post-vaccination) up to 6 months post-vaccination
Arm/Group | Menactra® Vaccine Group | Menjugate® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 1/61 | 2/62
Other Adverse Events (participants affected / at risk) | 50/61 | 40/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Vaccine Group (N=61) | Menjugate® Vaccine Group (N=62)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Rickets (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Vaccine Group (N=61) | Menjugate® Vaccine Group (N=62)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 6 (6)
Teething (Gastrointestinal disorders) | 13 (13) | 9 (10)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7)
Irritability (General disorders) | 4 (6) | 0 (0)
Pyrexia (General disorders) | 15 (20) | 14 (15)
Pyrexia (General disorders) | 30 (30) | 18 (18)
Irritability (Psychiatric disorders) | 50 (50) | 40 (40)
Injection site Tenderness (General disorders) | 36 (36) | 21 (21)
Injection site Erythema (General disorders) | 32 (32) | 23 (23)
Injection site Swelling (General disorders) | 18 (18) | 8 (8)
Somnolence (Nervous system disorders) | 31 (31) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 45 (45) | 24 (24)
Crying (Psychiatric disorders) | 31 (31) | 22 (22)
Nasopharyngitis (Infections and infestations) | 14 (19) | 8 (8)
Otitis media (Infections and infestations) | 7 (9) | 0 (0)
Roseola (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.